CLINICAL TRIAL: NCT02539329
Title: Characterization of Sensory Neuropathies Associated With Anti-FGFR3 Antibodies
Brief Title: Characterization of Anti-FGFR3 Antibodies
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1408060; 2014-A00636-41 (Other: ANSM)
Record Dates: First submitted 2015-07-31; First posted 2015-09-03 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Sensory Peripheral Neuropathy
Keywords: neuropathy; antibodies antiFGFR3; Biological diagnostic criteria
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for antibodies measure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient: Male or female patient aged 18 years with a clinically pure sensory peripheral neuropathy and positive for anti-FGFR3 antibodies. These patients will have Neurological assessment and Blood sample.
  Interventions: Other: Neurological assessment and Blood sample
- control: Male or female patient aged 18 years with a clinically pure sensory peripheral neuropathy and negative for anti-FGFR3 antibodies
  Interventions: Other: Neurological assessment and Blood sample

INTERVENTIONS:
Other: Neurological assessment and Blood sample — Neurological assessment (physical examination, electroneuromyography , International Prognostic Score (ISS), Overall Disability Scale (ODS), Rankin score) and 2 blood collection tubes for antibody screening

SUMMARY:
Sensory neuronopathies affect sensory neuron in the posterior spinal ganglion. They are responsible for pain, balance disorder (ataxia) and the use of hands. They depend on multiple etiologies. In a retrospective study, the investigators showed that the anti-FGFR3 antibody is a diagnostic marker of a subset of sensory neuronopathies. The investigators believe that other antibodies can be discovered in patients who remain seronegative changing.

However, the study is retrospective and only a small number of patients could be identified. Several points therefore need to be clarified or confirmed in a second prospective study.

DETAILED DESCRIPTION:
In and out patients evaluated for a sensory neuropathy meeting the inclusion and non-inclusion criteria will be proposed to enter the study

At inclusion the SSN diagnostic score is calculated and a blood sample is tested for anti-FGFR3 antibody.

Follow up: Patients positive for anti-FGFR3 antibodies will be followed and evaluated clinically and electrophysiologically at 1, 6 and 12 months. A blood sample is taken at 6 and 12 months.

A subgroup of patients negative for anti-FGFR3 antibodies will be randomly selected for evaluation at 1, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* A :Patients Male or female patient aged 18 years or more

Patients with a clinically pure sensory peripheral neuropathy including :

* idiopathic or dysimmune sensory neuronopathies
* idiopathic or dysimmune distal axonal sensory neuropathy
* sensory chronic inflammatory demyelinating polyradiculoneuropathy
* idiopathic or dysimmune small fiber neuropathies
* idiopathic or dysimmune trigeminal nerve neuropathy
* positive to antibodies anti-FGFR3

B :Controls Male or female patient aged 18 years or more

Patients with a clinically pure sensory peripheral neuropathy including :

* idiopathic or dysimmune sensory neuronopathies
* idiopathic or dysimmune distal axonal sensory neuropathy
* sensory chronic inflammatory demyelinating polyradiculoneuropathy
* idiopathic or dysimmune small fiber neuropathies
* idiopathic or dysimmune trigeminal nerve neuropathy
* negative to antibodies anti-FGFR3

Exclusion Criteria:

* -Motor or sensory-motor neuropathies
* Genetic, toxic, paraneoplasic neuropathies
* Diabetic Neuropathy.
* Neuropathy with Anti-MAG or anti-ganglioside IgM.
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient group : patient with clinically pure sensory peripheral neuropathy and positive for anti-FGFR3 antibodies Control group :clinically pure sensory peripheral neuropathy and negative for anti-FGFR3 antibodies
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Evolution of clinical and electrophysiological pattern of the neuropathy for patients with anti-FGFR3 antibodies (composite measure), | 6 months
  Score to the Overall Disability Scale Score (ODSS), the Rankin Score, the International PrognosticScore (ISS).

SECONDARY OUTCOMES:
Evolution of clinical and electrophysiological pattern of the neuropathy for patients with anti-FGFR3 antibodies (composite measure), | 12 months
  Score to the Overall Disability Scale Score (ODSS), the Rankin Score, the International PrognosticScore (ISS).
Description for patients with anti-FGFR3 antibodies of the immune context | 6 months
  Levels of Antibodies anti-FGFR3
Description for patients with anti-FGFR3 antibodies of the immune context | 12 months
  Levels of Antibodies anti-FGFR3
Patient evolution during one year for patients with anti-FGFR3 antibodies to a control group of sensory neuropathy without antibodies | 12 months
  Levels of Antibodies anti-FGFR3

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ANTOINE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (17):
- France (17):
  - CHU Bordeaux, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Chu Creteil, Créteil
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHRU de Nantes, Nantes
  - CHU de NICE, Nice
  - Hôpital BICETRE, Paris
  - Hopital Pitie Salpetriere, Paris
  - Fondation Rothschild, Paris
  - CHU Poitiers, Poitiers
  - CH Cornouailles, Quimper
  - CH Saint Denis - Hôpital Delafontaine, Saint-Denis
  - Chu Saint-Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg

REFERENCES:
- [Derived] Tholance Y, Moritz CP, Rosier C, Ferraud K, Lassabliere F, Reynaud-Federspiel E, Franca MC Jr, Martinez ARM, Camdessanche JP, Antoine JC; anti-FGFR3 antibody Study Group. Clinical characterisation of sensory neuropathy with anti-FGFR3 autoantibodies. J Neurol Neurosurg Psychiatry. 2020 Jan;91(1):49-57. doi: 10.1136/jnnp-2019-321849. Epub 2019 Nov 5. PMID 31690697